CLINICAL TRIAL: NCT00155246
Title: Phase 4 Study of the Efficacy of Pentoxifylline in Patients With Chronic Kidney Disease Receiving Angiotensin Receptor Blockade
Brief Title: Efficacy of Pentoxifylline on Chronic Kidney Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Shuei-Liong Lin/Attending Physician, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 930202
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2010-01-29 (Estimated); Status verified 2010-01

CONDITIONS: Chronic Kidney Disease
Keywords: CKD, pentoxifylline
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Pentoxifylline; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: pentoxifylline (drug)

SUMMARY:
To study whether pentoxifylline has additive renoprotective effect in patients taking ARB

DETAILED DESCRIPTION:
In patients with CKD and serum creatinine 1.3~6.0 md/gl, having taken losartan 100 mg/day for at least 3 months, with stable renal function, will be recruited to a randomized open-label trial. Patients taking pentoxifylline or not will be compared for their spot urinary proteinuria, estimated glomerular filtration, spot urine tumor necrosis factor-α/creatinine ratio, spot urine monocyte-chemoattractant protein-1/creatinine, and aldosterone concentration between groups in a 2-year study. Add-on pentoxifylline in control group in the same dose as in treat group will be performed to observe the renoprotective effect if any protective potential is demonstrated in the end of maintenance 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease with serum creatinine 1.3~6.0 mg/dl

Exclusion Criteria:

* History of allergy to pentoxifylline
* Females are nursing or pregnant
* Obstructive uropathy
* Unable to stop chronic immunosuppressive therapy, NSAID
* Congestive heart failure (New York Heart Association functional class III or IV)
* Unstable angina, myocardial infarction, coronary artery bypass graft surgery, percutaneous coronary intervention, within the past 6 months prior to signing the informed consent form
* Cerebral hemorrhage within the past 6 months prior to signing the informed consent form
* Retinal hemorrhage within the past 6 months prior to signing the informed consent form
* Known or suspected secondary hypertension (e.g., primary aldosteronism, renovascular hypertension, pheochromocytoma)
* Severe uncontrolled hypertension with SBP > 220 mmHg and/or DBP > 115 mmHg
* Hepatic dysfunction as defined by the following laboratory parameters: ALT or AST > 2 times the upper limit of the normal range
* Biliary obstructive disorders (e.g. cholestasis)
* Active malignancy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-07; Primary Completion 2006-07 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
spot urinary proteinuria between groups

SECONDARY OUTCOMES:
estimated glomerular filtration, spot urine tumor necrosis factor-α/creatinine ratio, spot urine monocyte-chemoattractant protein-1/creatinine, and aldosterone concentration between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Tun-Jun Tsai, MD, PhD, Principal Investigator — National Taiwan University Hosptial
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Natale P, Mooi PK, Palmer SC, Cross NB, Cooper TE, Webster AC, Masson P, Craig JC, Strippoli GF. Antihypertensive treatment for kidney transplant recipients. Cochrane Database Syst Rev. 2024 Jul 31;7(7):CD003598. doi: 10.1002/14651858.CD003598.pub3. PMID 39082471